CLINICAL TRIAL: NCT07145905
Title: A Prospective, Open-label, Multicenter, Interventional Study, to Evaluate Safety and Efficacy of TCRM in the Treatment of the Cheek Area Including Fine Lines: SPARKS
Brief Title: TCRM for Correction of Cheek Including Fine Lines
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEO-TCRM-2204
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Skin Aging; Cheek Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCRM (Experimental): Treatments performed in this study include:
  * An initial injection at V1 during which subjects will be injected with TCRM in the cheek area.
  * An optional touch-up injection 4 weeks after the initial injection (at V2).
  Interventions: Device: TCRM

INTERVENTIONS:
Device: TCRM — N=128

SUMMARY:
The purpose of this clinical study is to evaluate benefits and risks of injecting TCRM in the cheek including fine lines. The goal is to show that treatment with TCRM will result in correcting the cheek area including the fine lines at 4 weeks after last treatment (initial injection or touch up) on subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects over 18 years old seeking correction of the cheek area including fine lines.
* Subject scored grade 1 to 3 on the CFLDS.
* For women: not pregnant, not breast feeding
* Female subjects of childbearing potential must have a negative UPT and practice a reliable method of contraception throughout the study.
* Willing to abstain from facial aesthetic procedures/therapies that could interfere with study evaluations
* Able to follow study instructions and complete all required visits.
* Having given its signed informed consent.

Exclusion Criteria:

* Known hypersensitivity or previous allergic reaction to any component of the study devices
* Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, or history of anaphylactic shock.
* History of active chronic debilitating systemic disease that, in the opinion of the investigator, would make the subject a poor candidate in the study.
* Subject exhibits any physical attribute that may prevent assessment or treatment of the cheek area including fine lines as judged by the PI
* Clinically significant alcohol or drug abuse.
* Subject has received any investigational product within 90 days prior to Visit 1 or planning to participate in another investigation during the course of the study.
* Subject has unstable weight, as judged by the PI.
* Subject has no teeth or misses significant portion of dentition that changes the face appearance (subjects with dentures sufficiently replacing missing natural teeth are allowed).
* Subject under guardianship/tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the efficacy of TCRM in the treatment of the cheek area including fine lines at 4 weeks after last injection (initial injection or touch up) using Global Aesthetic Improvement Scale (GAIS) as assessed by both subject and PI. | 4 weeks after last injection
  The Global Aesthetic Improvement (GAI) is a subjective, balanced, 5-point dynamic scale assessing cosmetic improvement.
  Possible scores range from "much improved", "improved", "no change", "worse", to "much worse"

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico Lajo Rosso, Madrid, Spain